CLINICAL TRIAL: NCT01019980
Title: A Comparative Double Blind, Double Dummy, Randomized Study on the Effectiveness of Diclofenac Potassium vs. Acetaminophen in Febrile Children With Acute Upper Respiratory Tract Infections
Brief Title: Efficacy of Diclofenac Potassium Versus Acetaminophen in Febrile Children With Acute Upper Respiratory Tract Infections
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Placebo - Active Drug Not Available. No patients received drug. There are no study results to disclose.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVOL458AVE02
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-10

CONDITIONS: Fever
Keywords: Antipyretics; fever; diclofenac; acetaminophen; children; acute upper respiratory tract infections
MeSH Terms: conditions — Fever | interventions — Diclofenac; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Diclofenac potassium (Experimental)
  Interventions: Drug: Diclofenac potassium
- Acetaminophen (Active Comparator)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Diclofenac potassium — Diclofenac potassium
  Arms: Diclofenac potassium
Drug: Acetaminophen — Acetaminophen
  Arms: Acetaminophen

SUMMARY:
The purpose of this study is to assess if a single dose of Diclofenac potassium (0.5 mg/kg) is more or as effective as a single dose of Acetaminophen (10 mg/kg) in the reduction of fever during 2 hours, in the treatment of febrile children with acute upper respiratory infections.

This is a comparative double blind, double dummy, randomized study on the effectiveness of Diclofenac potassium versus Acetaminophen in febrile children with acute upper respiratory tract infections. The patient will be randomized to either group: Group A (Diclofenac potassium (0.5 mg/kg) or Group B (Acetaminophen (10 mg/kg)). A Health Care Professional trained will measure the temperature during 2 hours. During the study period, parents or legal representatives will be invited to fill a survey about the habits and knowledge regarding fever management at home.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, aged 2 to 6 years presenting tympanic temperature ≥ 38.5 ° C and no greater than 39.5° C, associated with acute upper respiratory tract infections
* Parents or legal representatives who have provided written informed consent and provided a phone number for the call at end of study

Exclusion Criteria:

* History of hypersensitivity to any drugs or excipients of the study
* Any medication, surgical, or medical condition, which might significantly alter the absorption, distribution, metabolism, or excretion of medications
* Background or suspected hematological disorders, febrile seizures, asthma, peptic ulcer or gastrointestinal bleeding
* Neurological and hemodynamics disorders
* Evidence of liver or kidney impairment or heart failure
* Patients who have received previous treatment with antipyretics; acetaminophen (up to 4 hrs), NSAIDs (up to 6 hrs) or antibiotic therapy (at least 12 hours)
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at risk

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Venezuela (2):
  - Hospital de niños "J. M. de los Rios", Distrito Metropolitano, Caracas
  - Ciudad Hospitalaria Enrique Tejera, Valencia, Estado Carabobo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants entered the study but did not receive drug because drug was not available in the region. The study was then terminated.
Groups:
- Diclofenac Potassium: This study was cancelled. Two patients were enrolled, but neither received drug as it was not available in the region
- Acetaminophen: This study was cancelled. No patients were enrolled in this group.
Period: Overall Study
Arm/Group | Diclofenac Potassium | Acetaminophen
Started | 2 (2 patients entered study but did not receive any drug since it was not available in the region.) | 0
Discontinued | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Drug not available. | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Potassium | Acetaminophen | Total
Number analyzed (Participants) | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — This study was cancelled. Two patients were enrolled, but neither received drug as it was not available in the region
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Reduction of Temperature
Time Frame: 2 hours
Arm/Group | Diclofenac Potassium | Acetaminophen
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Reach a Reduction of Temperature as 0.5 and 1 °C
Time Frame: 2 hours
Reporting Status: Not Posted

3. Secondary Outcome: Time With a Temperature ≤ 38,4 °C in a Period of 6 Hours
Time Frame: 6 hours
Reporting Status: Not Posted

4. Secondary Outcome: Safety of Diclofenac Potassium Therapy in the Study Period
Time Frame: 6 hours
Reporting Status: Not Posted

5. Secondary Outcome: The Level of Knowledge That Parents or Legal Representatives Have on the Treatment of Fever
Time Frame: 2 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Diclofenac Potassium | Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was cancelled. Two patients were enrolled, but neither received drug as it was not available in the region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.